

## TÜRKİYE CUMHURİYETİ İSTANBUL AYDIN ÜNİVERSİTESİ

## THE REPUBLIC OF TÜRKİYE ISTANBUL AYDIN UNIVERSITY

T.C. İSTANBÜL 2005 IN ÖYİVERSİTESİ GİRİŞİMSEL OLMAYAN KLİNİK XRAŞTIŞİM ALAR ETİK KURULU KARARI

ARAŞTIRMANIN AÇIK ADI Kronik Bel Ağrılı Kadın Hastalarda Konvansiyonel Tedaviye Ek Olarak Uygulanan Dinamik Nöromusküler Stabilizasyon Egzersizlerinin Fonksiyonel Kapasiteye, Core Stabilizasyon Kaslarının Kuvvetine ve Dengeye Etkisi

| BAȘVURU BİLGİLERİ | KOORDİNATÖR/SORUMLU<br>ARAŞTIRMACI<br>UNVANI/ADI/SOYADI | Dr. Öğr. Üyesi | Gözde Başbu | ğ | |
|---|---|---|---|---|---|
| | KOORDİNATÖR/SORUMLU<br>ARAŞTIRMACININ UZMANLIK<br>ALANI | Fizyoterapi ve Rehabilitasyon | | | |
| | KOORDİNATÖR/SORUMLU<br>ARAŞTIRMACININ BULUNDUĞU<br>MERKEZ | Sağlık Bilimleri Fakültesi | | | |
| | VARSA DESTEKLEYİCİ | - | | | |
| | VARSA DESTEKLEYİCİNİN<br>YASAL TEMSİLCİSİ | - | | | |
| | ARAŞTIRMANIN TİPİ | Gözlemsel Çalışma | | | |
| | ARAŞTIRMAYA KATILAN<br>MERKEZLER | TEK<br>MERKEZ | ÇOK<br>MERKEZLİ | ULUSAL<br>X | ULUSLAR-<br>ARASI |

| Belge Adı | Tarihi | Dili |
|---|---|---|
| ARAŞTIRMA PROTOKOLÜ | 16.01.2025 | Türkçe X İngilizce Diğer |
| BİLGİLENDİRİLMİŞ GÖNÜLLÜ<br>OLUR FORMU | 16.01.2025 | Türkçe X İngilizce ☐ Diğer ☐ |
| OLGU RAPOR FORMU | 16.01.2025 | Türkçe X İngilizce Diğer Diğer |
| ARŞİV MATERYALİ KULLANIMI<br>İÇİN TAAHHÜTNAME | - | |
| Belge Adı | | Açıklama |
| DİĞER: | 16.01.2025 | Dilekçe (Ön Bilgi Formu), Beyan Formu,<br>Çalışma Akış Şeması, Helsinki Bildirgesi,<br>Araştırma Bütçe Formu, Kurum İzni, İKU<br>Bilgilendirme Belgesi, Özgeçmişler, Literatürler |
| Karar No: 28/2025 | Tarih: 12.0 | )2.2025 |
| | ARAŞTIRMA PROTOKOLÜ BİLGİLENDİRİLMİŞ GÖNÜLLÜ OLUR FORMU OLGU RAPOR FORMU ARŞİV MATERYALİ KULLANIMI İÇİN TAAHHÜTNAME Belge Adı DİĞER: | ARAŞTIRMA PROTOKOLÜ BİLGİLENDİRİLMİŞ GÖNÜLLÜ OLUR FORMU OLGU RAPOR FORMU ARŞİV MATERYALİ KULLANIMI İÇİN TAAHHÜTNAME Belge Adı DİĞER: 16.01.2025 |

Sayın, Dr. Öğr. Üyesi Gözde BAŞBUĞ

İstanbul Aydın Üniversitesi Girişimsel Olmayan Klinik Araştırmalar Etik Kurulu'nun 12.02.2025 tarihinde yapılan olağan toplantısında danışmanlığını yürüttüğünüz "Safiye Esin" isimli öğrencinize ait "Kronik Bel Ağrılı Kadın Hastalarda Konvansiyonel Tedaviye Ek Olarak Uygulanan Dinamik Nöromusküler Stabilizasyon Egzersizlerinin Fonksiyonel Kapasiteye, Core Stabilizasyon Kaslarının Kuvvetine ve Dengeye Etkisi" konulu yüksek lisans tez araştırmanız ile ilgili alınan 28/2025 no'lu karar gereği; başvuru dosyanız ile ilgili belgeler araştırmanın gerekçe, amaç, yaklaşım ve yöntemleri dikkate alınarak incelenerek etik ve bilimsel yönden uygun olduğuna "Oy birliği" ile karar verilmiştir.

Bilgilerinize sunarım.

Etik Kurul Başkanının Unvanı/Adı/Soyadı: Prof. Dr. Erman/Bülent TUNCER

KARAR BİLGİLERİ

## İSTANBUL AYDIN ÜNİVERSİTESİ GİRİŞİMSEL OLMAYAN KLİNİK ARAŞTIRMALAR ETİK KURULU

BAŞKANIN UNVANI / ADI / SOYADI:

Prof. Dr. Erman Bülent TUNCER

| Unvanı/Adı/Soyadı | Uzmanlık<br>Alanı | Birimi | Araştırma<br>ile ilişki | | Katılım | | İmza |
|---|---|---|---|---|---|---|---|
| Prof. Dr. Erman<br>Bülent TUNCER | Protetik Diş<br>Tedavisi | Diş Hekimliği<br>Fakültesi | Е | H<br>X | Е | Н | |
| Prof. Dr. Hatice Aysel<br>ALTAN | Anesteziyoloji<br>ve<br>Reanimasyon | Sağlık Hizmetleri<br>Meslek<br>Yüksekokulu | Е | H<br>X | Е | Н | Cupersen |
| Doç. Dr. Türkiz<br>VERİMER | Farmakoloji | Sağlık Hizmetleri<br>Meslek<br>Yüksekokulu | Е | H<br>X | Е | Н | 7.125. |
| Prof. Dr. Hafize<br>SEZER | Biyoistatistik | Tıp Fakültesi | Е | H<br>X | Е | Н | lane |
| Prof. Dr. Demet<br>Funda BAŞ | Nöroloji | Tıp Fakültesi | Е | H<br>X | Е | Н | MM. |
| Doç. Dr. Didem<br>ÖNER ÖZDAŞ | Endodonti | Diş Hekimliği<br>Fakültesi | Е | H<br>X | Е | Н | - functions |
| Doç. Dr. Hasret<br>AYYILDIZ CİVAN | Çocuk Sağlığı<br>ve<br>Hastalıkları | Tıp Fakültesi | Е | H<br>X | Е | Н | She |
| Prof. Dr. Ebru<br>CEYLAN | Hukuk | Hukuk Fakültesi | Е | H<br>X | Е | Н | Ebulyton |
| Dr. Öğr. Üyesi Özge<br>YILMAZLI | Tıbbi<br>Mikrobiyoloji | Tıp Fakültesi | Е | H<br>X | Е | Н | |
| Dr. Öğr. Üyesi<br>Hüseyin KAZAN | Gazetecilik | İletişinı Fakültesi | Е | H<br>X | Е | Н | (Ching) |
| Doç. Dr. Dilek<br>YILDIRIM | Hemşirelik | Sağlık Bilimleri<br>Fakültesi | Е | H<br>X | Е | Н | DYM |

Etik Kurul Başkanının

Unvanı/Adı/Soyadı: Prof. Dr. Erman Bülent TUNCER

İmza:

Not: Etik kurul başkanı, imzasının yer almadığı her sayfaya imza atmalıdır.